CLINICAL TRIAL: NCT02681575
Title: Meta-cognitive Functional Intervention for Adults (Cog-Fun - A) With Attention Deficit Hyperactivity Disorder (ADHD): A Pilot Efficacy Study
Brief Title: Meta-cognitive Functional Intervention for Adults With ADHD: A Pilot Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0658-15-HMO
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2016-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cog-Fun A (Experimental): Metacognitive-Functional occupational therapy intervention (Cog-Fun - A) includes enhancing self awareness in occupational context, acquiring executive strategies and skills and implementation across multiple occupational domains.
  Interventions: Behavioral: Cog-Fun - A

INTERVENTIONS:
Behavioral: Cog-Fun - A — Meta-cognitive functional intervention for improved self management in adults with ADHD

SUMMARY:
The purpose of this study is to examine the initial efficacy of a psycho-social, metacognitive-functional intervention for Adults (Cog-Fun - A) with Attention Deficit Hyperactivity Disorder (ADHD).

It is hypothesized that participants in the Cog-Fun - A intervention will demonstrate improvements in measures of executive functioning, occupational performance and quality of life.

DETAILED DESCRIPTION:
The Cog-Fun - A is a structured occupational therapy intervention for promoting self management in adults with ADHD. The protocol comprises three central treatment modules: Adaptive self awareness, executive strategies and skill implementation and multi-context transfer of strategies and skills.

The intervention is administered by occupational therapists on an individual basis, once a week, over 3-4 months.

20 participants will be recruited through community advertising. Sample size was determined based on expected moderate effect sizes. Data will be collected at the onset and completion of the intervention. Data will be analysed using quantitative and qualitative methods.

Adverse events if occur will be reported to supervising psychiatrist and the Helsinki Committee.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosed by certified medical practitioner
* Adult ADHD Self Report Scale (ASRS) score above cutoff
* BRIEF-A score above cutoff

Exclusion Criteria:

* Diagnoses of severe neurological or psychiatric health condition.
* Instability in pharmacological treatment
* Brief Symptom Inventory (BSI) above cutoff according to Israeli adult norms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Behavioral Ratings of Executive Functions - Adult version (BRIEF-A) | 3-4 months
  Self rating questionnaire targeting executive functions in daily life

SECONDARY OUTCOMES:
Adult ADHD Quality of Life Scale (AaQoL) | 3-4 months
  Self rating questionnaire targeting the impact of ADHD on Life Productivity, Psychological Health, Relationships and Life outlook
Canadian Occupational Performance Measure | 3-4 months
  structured interview administered by occupational therapist

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bonne, MD, Principal Investigator — HMO
Locations (1):
- Hadassah Medical Organization, Mount Scopus, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided